CLINICAL TRIAL: NCT04788082
Title: Clinical Impact of Rapid Prototyping 3D Models of Congenital Heart Disease on Surgical Management
Brief Title: Clinical Impact of Rapid Prototyping 3D Models for Surgical Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollments
Sponsor: Children's National Research Institute (Other)
Collaborators: Phoenix Children's Hospital (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Laura Olivieri, Cardiologist, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-090
Record Dates: First submitted 2017-08-29; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Double Outlet Right Ventricle; Transposition of the Great Arteries; Truncus Arteriosus; Congenitally Corrected Transposition of the Great Arteries
Keywords: 3D Printing; Rapid prototpying
MeSH Terms: conditions — Double Outlet Right Ventricle; Transposition of Great Vessels; Truncus Arteriosus, Persistent; Congenitally Corrected Transposition of the Great Arteries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care (not involving 3D printing)
- 3D Model (Experimental): 3D printed models (at least one rigid blood volume model and one flexible shell model) will be used for surgical planning.
  Interventions: Diagnostic Test: 3D Printed Heart Model

INTERVENTIONS:
Diagnostic Test: 3D Printed Heart Model — Prior to surgical intervention, the surgeon will be exposed to clinically-indicated images and a patient-specific 3D printed model of the subject's heart anatomy.
  Other Names: Rapid Prototyped Heart Model
  Arms: 3D Model

SUMMARY:
Patient-specific, 3D printed models have been utilized in preoperative planning for many years. Among researchers and clinicians, there is a perception that preoperative exposure to 3D printed models, derived from patient images (CT or MRI), aid in procedural planning. 3D printed models for heart surgery have the potential to improve a clinician's preparedness and therefore may reduce surgically-related morbidity and mortality. This randomized clinical trial aims to evaluate whether pre-procedural planning of surgeons exposed to a patient-specific 3D printed heart model will decrease cardiopulmonary bypass time, morbidity, and mortality.

DETAILED DESCRIPTION:
3D imaging and rapid prototyping 3D printing technology have advanced to the point where it is feasible to marry the two to produce a patient-matched and accurate 3D model of congenital heart defects. The production of a 3D model of the heart may be particularly useful in anticipation of surgery such that the operator can plan and visualize the surgery prior to the surgical date with a physical heart he or she can manipulate in their hands.

Preliminary studies demonstrate potential for clinical impact of 3D models on patient care and patient outcomes. 3D models have long been shown to enhance education and communication of anatomy. In 2008 Kim et al reviewed 3D printed models as an emerging technology in management of congenital heart disease, and also suggests that physical models may also help enhance patients and physicians' understanding of congenital heart disease. Our group has also published on the clinical and educational value of these 3D heart models. To date, no systematic trial identifying the value of 3D models on procedural planning has been published.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects undergoing primary complex two-ventricle repair of congenital heart defect, including but not limited to:

  1. double outlet right ventricle (DORV),
  2. transposition of the great arteries with ventricular septal defect and pulmonary stenosis (TGA/VSD/PS),
  3. truncus arteriosus with ventricular septal defect (TA/VSD)
  4. congenitally corrected transposition of the arteries with pulmonary stenosis (CCTGA/PS).
* Patient who will undergo preoperative cardiac MR or cardiac CT imaging

  a. Images will be validated by the IRC prior to inclusion
* Written informed consent (and assent when applicable) and HIPAA authorization obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Complex defects involving atrioventricular valve anomalies

  1. complete or transitional atrioventricular canal
  2. double inlet left ventricle
  3. tricuspid atresia
  4. mitral atresia
* Defects with valve dysfunction requiring an extensive valvuloplasty
* Patients with a contraindication to MRI scanning will be excluded unless they are referred for a cardiac CT per clinical standard of practice. These contraindications include patients with the following devices:

  1. Central nervous system aneurysm clips
  2. Implanted neural stimulator
  3. Implanted cardiac pacemaker or defibrillator which are not MR safe or MR conditional according to the manufacturer
  4. Cochlear implant
  5. Ocular foreign body (e.g. metal shavings)
  6. Implanted Insulin pump
  7. Metal shrapnel or bullet.
  8. Any contraindications to receiving IV gadolinium contrast, determined clinically
* Subjects where MRI or CT images are acquired more than six months prior to the scheduled surgical date
* Subjects where date of scan to date of surgery is less than 10 calendar days
* Subjects where MRI or CT reconstruction is limited due to poor image acquisition as solely determined by the Image Reconstruction Center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time under cardiopulmonary bypass | peri-operative

SECONDARY OUTCOMES:
Mortality | Up to 30 days post-operative
Intraoperative death or intraprocedural death | peri-operative
Unexpected Cardiac arrest during or following procedure | From surgical date through 30 days post-operative
Bleeding, Requiring reoperation | From surgical date through 30 days post-operative
Sternum left open, Unplanned | From surgical date through 30 days post-operative
Unplanned cardiac reoperation | From surgical date through 30 days post-operative
Unplanned non-cardiac reoperation | From surgical date through 30 days post-operative
Mechanical circulatory support (IABP, VAD, ECMO, or CPS) | From surgical date through 30 days post-operative
  Answer "yes"/"no"
Arrhythmia necessitating pacemaker, Permanent pacemaker | From surgical date through 30 days post-operative
Renal failure (discharge dialysis) | From surgical date through 30 days post-operative
  acute renal failure, Acute renal failure requiring dialysis at the time of hospital discharge
Renal failure (temporary dialysis) | From surgical date through 30 days post-operative
  acute renal failure, Acute renal failure requiring temporary dialysis with the need for dialysis not present at hospital discharge
Renal failure (hemofiltration) | From surgical date through 30 days post-operative
  acute renal failure, Acute renal failure requiring temporary hemofiltration with the need for dialysis not present at hospital discharge
Sepsis | From surgical date through 30 days post-operative
  Sepsis (following Society of Thoracic Surgery definition)
Seizure | From surgical date through 30 days post-operative
  Seizure (following Society of Thoracic Surgery definition)
Stroke | From surgical date through 30 days post-operative
  Stroke (following Society of Thoracic Surgery definition)
Vocal cord dysfunction (possible recurrent laryngeal nerve injury) | From surgical date through 30 days post-operative
Other operative/procedural complication | From surgical date through 30 days post-operative
  Other operative/procedural complication (following Society of Thoracic Surgery definition)
Technology Assessment | Preop, Periop, and up to 30 days a
  A survey will be given to the surgeons assessing technology acceptance of the 3D printed heart models

CONTACTS AND LOCATIONS:
Overall Officials: Laura Olivieri, MD, Principal Investigator — Children's National Research Institute; Stephen Pophal, MD, Principal Investigator — Phoenix Children's Hospital; Yoav Dori, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardoen B, Demeulemeester E, Beliën J. Operating room planning and scheduling: A literature review. European Journal of Operational Research 201(3): 921-932, 2010.
- [Background] Costello JP, Olivieri LJ, Krieger A, Thabit O, Marshall MB, Yoo SJ, Kim PC, Jonas RA, Nath DS. Utilizing Three-Dimensional Printing Technology to Assess the Feasibility of High-Fidelity Synthetic Ventricular Septal Defect Models for Simulation in Medical Education. World J Pediatr Congenit Heart Surg. 2014 Jul;5(3):421-6. doi: 10.1177/2150135114528721. PMID 24958045
- [Background] Costello JP, Olivieri LJ, Su L, Krieger A, Alfares F, Thabit O, Marshall MB, Yoo SJ, Kim PC, Jonas RA, Nath DS. Incorporating three-dimensional printing into a simulation-based congenital heart disease and critical care training curriculum for resident physicians. Congenit Heart Dis. 2015 Mar-Apr;10(2):185-90. doi: 10.1111/chd.12238. Epub 2014 Nov 11. PMID 25385353
- [Background] Cui X, Boland T, D'Lima DD, Lotz MK. Thermal inkjet printing in tissue engineering and regenerative medicine. Recent Pat Drug Deliv Formul. 2012 Aug;6(2):149-55. doi: 10.2174/187221112800672949. PMID 22436025
- [Background] Davis FD, Bagozzi RP, Warshaw PR. User Acceptance of Computer Technology: A Comparison of Two Theoretical Models. Management Science 35(8): 982-1003, 1989.
- [Background] Dexter F, Macario A. Changing allocations of operating room time from a system based on historical utilization to one where the aim is to schedule as many surgical cases as possible. Anesth Analg. 2002 May;94(5):1272-9, table of contents. doi: 10.1097/00000539-200205000-00042. PMID 11973204
- [Background] Does RJMM, Vermaat TMB, Verver JPS, Bisgaard S, Van Den Heuvel J. Reducing Start Time Delays in Operating Rooms. Journal of Quality Technology 41(1): 95-109, 2009.
- [Background] Ejaz F, Ryan J, Henriksen M, Stomski L, Feith M, Osborn M, Pophal S, Richardson R, Frakes D. Color-coded patient-specific physical models of congenital heart disease. Rapid Prototyping Journal 20(4): 336-343, 2014.
- [Background] Gelijns AC, Moskowitz AJ, Acker MA, Argenziano M, Geller NL, Puskas JD, Perrault LP, Smith PK, Kron IL, Michler RE, Miller MA, Gardner TJ, Ascheim DD, Ailawadi G, Lackner P, Goldsmith LA, Robichaud S, Miller RA, Rose EA, Ferguson TB Jr, Horvath KA, Moquete EG, Parides MK, Bagiella E, O'Gara PT, Blackstone EH; Cardiothoracic Surgical Trials Network (CTSN). Management practices and major infections after cardiac surgery. J Am Coll Cardiol. 2014 Jul 29;64(4):372-81. doi: 10.1016/j.jacc.2014.04.052. PMID 25060372
- [Background] Hu A, Wilson T, Ladak H, Haase P, Doyle P, Fung K. Evaluation of a three-dimensional educational computer model of the larynx: voicing a new direction. J Otolaryngol Head Neck Surg. 2010 Jun;39(3):315-22. PMID 20470679
- [Background] Kim MS, Hansgen AR, Wink O, Quaife RA, Carroll JD. Rapid prototyping: a new tool in understanding and treating structural heart disease. Circulation. 2008 May 6;117(18):2388-94. doi: 10.1161/CIRCULATIONAHA.107.740977. PMID 18458180
- [Background] King WR, He J. A meta-analysis of the technology acceptance model. Information & Management 43(6): 740-755, 2006.
- [Background] Kutty S, Graney BA, Khoo NS, Li L, Polak A, Gribben P, Hammel JM, Smallhorn JF, Danford DA. Serial assessment of right ventricular volume and function in surgically palliated hypoplastic left heart syndrome using real-time transthoracic three-dimensional echocardiography. J Am Soc Echocardiogr. 2012 Jun;25(6):682-9. doi: 10.1016/j.echo.2012.02.008. Epub 2012 Mar 14. PMID 22421029
- [Background] Lang RM, Badano LP, Tsang W, Adams DH, Agricola E, Buck T, Faletra FF, Franke A, Hung J, de Isla LP, Kamp O, Kasprzak JD, Lancellotti P, Marwick TH, McCulloch ML, Monaghan MJ, Nihoyannopoulos P, Pandian NG, Pellikka PA, Pepi M, Roberson DA, Shernan SK, Shirali GS, Sugeng L, Ten Cate FJ, Vannan MA, Zamorano JL, Zoghbi WA; American Society of Echocardiography; European Association of Echocardiography. EAE/ASE recommendations for image acquisition and display using three-dimensional echocardiography. J Am Soc Echocardiogr. 2012 Jan;25(1):3-46. doi: 10.1016/j.echo.2011.11.010. No abstract available. PMID 22183020
- [Background] Mavroudis C, Backer C, Idriss RF. Pediatric Cardiac Surgery, 4 edition. Hoboken, NJ, Wiley-Blackwell, 2012.
- [Background] Moreno Cegarra JL, Cegarra Navarro JG, Córdoba Pachón JR. Applying the technology acceptance model to a Spanish City Hall. International Journal of Information Management 34(4): 437-445, 2014.
- [Background] Mottl-Link S, Hubler M, Kuhne T, Rietdorf U, Krueger JJ, Schnackenburg B, De Simone R, Berger F, Juraszek A, Meinzer HP, Karck M, Hetzer R, Wolf I. Physical models aiding in complex congenital heart surgery. Ann Thorac Surg. 2008 Jul;86(1):273-7. doi: 10.1016/j.athoracsur.2007.06.001. PMID 18573436
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Olivieri L, Krieger A, Chen MY, Kim P, Kanter JP. 3D heart model guides complex stent angioplasty of pulmonary venous baffle obstruction in a Mustard repair of D-TGA. Int J Cardiol. 2014 Mar 15;172(2):e297-8. doi: 10.1016/j.ijcard.2013.12.192. Epub 2014 Jan 8. No abstract available. PMID 24447757
- [Background] Ryan JR, Moe TG, Richardson R, Frakes DH, Nigro JJ, Pophal S. A novel approach to neonatal management of tetralogy of Fallot, with pulmonary atresia, and multiple aortopulmonary collaterals. JACC Cardiovasc Imaging. 2015 Jan;8(1):103-104. doi: 10.1016/j.jcmg.2014.04.030. Epub 2014 Nov 12. No abstract available. PMID 25457761
- [Background] Sodian R, Weber S, Markert M, Rassoulian D, Kaczmarek I, Lueth TC, Reichart B, Daebritz S. Stereolithographic models for surgical planning in congenital heart surgery. Ann Thorac Surg. 2007 May;83(5):1854-7. doi: 10.1016/j.athoracsur.2006.12.004. PMID 17462413
- [Background] Weidenbach M, Razek V, Wild F, Khambadkone S, Berlage T, Janousek J, Marek J. Simulation of congenital heart defects: a novel way of training in echocardiography. Heart. 2009 Apr;95(8):636-41. doi: 10.1136/hrt.2008.156919. Epub 2009 Jan 8. PMID 19131439
- [Background] Wypij D, Newburger JW, Rappaport LA, duPlessis AJ, Jonas RA, Wernovsky G, Lin M, Bellinger DC. The effect of duration of deep hypothermic circulatory arrest in infant heart surgery on late neurodevelopment: the Boston Circulatory Arrest Trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1397-403. doi: 10.1016/s0022-5223(03)00940-1. PMID 14666011
- [Background] Yarbrough AK, Smith TB. Technology acceptance among physicians: a new take on TAM. Med Care Res Rev. 2007 Dec;64(6):650-72. doi: 10.1177/1077558707305942. Epub 2007 Aug 23. PMID 17717378
- See also: Phoenix Children's Hospital's 3D Print Lab — http://Cardiac3DPrintLab.com
- See also: Children's National Medical Center — http://childrensnational.org/